CLINICAL TRIAL: NCT07065188
Title: Effect of Pain Vigilance on Pain Catastrophizing, Bladder-Bowel Function and Sexual Life: A Comparative Study of Before-After Vaginal Surgery
Brief Title: Effect of Pain Vigilance on Pain, Bladder-Bowel Function and Sexual Life
Status: Not yet recruiting | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Semiha Yenişehir, PT, PhD, Assist. Prof. Dr., Ordu University
Other Study IDs: 2025 06/254
Record Dates: First submitted 2025-06-30; First posted 2025-07-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Vaginal Surgery
Keywords: Vaginal surgery; pain vigilance; sexual function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study to investigate the effect of preoperative pain hypervigilance on postoperative pain, bladder-bowel symptoms and sexual life after vaginal surgery and to compare these parameters before and after surgery. Pain vigilance (Pain Vigilance and Awareness Questionnaire-PVAQ), pain catastrophizing (Pain Catastrophizing Scale-PCS), bladder-bowel function (Australian Pelvic Floor Questionnaire-APFQ), and sexual function (Female Sexual Function Index (FSFI)) of women were recorded before and after surgery. Visual analogue scales were used to assess the postoperative pain intensity.

DETAILED DESCRIPTION:
Hypervigilance is the state of being consciously alert to external stimuli. Specific attention to pain or other somatosensory stimuli is defined as "specific hypervigilance". Hypervigilance is a strong indicator of subjective acute postoperative pain and contributes significantly to the prediction of post-operative pain. A cautious bias toward positive preoperative stimuli may predispose patients to postoperative pain, indicating a maladaptive coping method. Pain-related disability occurs in patients with a high level of pain hypervigilance before surgery. Urinary and bowel functions are impaired after vaginal surgery and bladder-bowel dysfunction is observed. Sexual function is also affected positively or negatively after vaginal surgery. The causes of sexual dysfunction after vaginal surgery are classified as organic, emotional and psychological. Decreased pelvic blood flow may cause vaginal dryness and dyspareunia by causing vaginal smooth muscle fibrosis.

This study was planned to evaluate the effect of preoperative pain hypervigilance on post-operative pain, bladder-bowel symptoms and sexual life in women undergoing vaginal surgery and to compare these parameters before and after surgery. Physical and sociodemographic, obstetric and clinical characteristics will be recorded. Pain, bladder-bowel and sexual function will be evaluated before and after surgery. The pain trigger status of the subjects will be assessed with the PVAQ, the degree to which they catastrophize pain will be assessed with the PCS and their sexual function will be assessed with the FSFI . The AOFQ will be used to assess bladder-bowel function. Postoperative pain intensity during urination and defecation will be evaluated with Visual Analog Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18-40.
* Being able to read and write Turkish.
* Have undergone vaginal surgery.

Exclusion Criteria:

* Presence of any confounding condition in post-operative pain severity (patients with a history of chronic pelvic pain and/or endometriosis or pelvic inflammatory disease),
* Having conditions in which sexual activity is contraindicated and should be restricted (genital infection, etc.),
* Vulvovaginal infection,
* Having a neurological disease,
* Having visual, auditory, and cognitive problems that may prevent participation in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Have undergone vaginal surgery
Sampling Method: Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain Vigilance and Awareness Questionnaire | Before and first day of after surgery (first postoperative day)
  The Turkish version of the PVAQ will be used to measure alertness to pain and pain awareness. In the 16-item Likert-type questionnaire, "never" equals 0, "rarely" equals 1, "sometimes" equals 4 and "always" equals 5 points. Items 8 and 16 of the questionnaire are reverse scored. The lowest score is 0 and the highest score is 80. A higher score indicates more pain awareness.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | Before and first day of after surgery (first postoperative day)
  This scale was developed to measure the exaggerated negative mental reaction of individuals to existing or anticipated painful experiences and the extent to which they catastrophize pain. The validity and reliability of the Turkish version of the scale was demonstrated. It consists of 13 items, and each item is scored as never=0, slightly=1, moderately=2, greatly=3 and always=4. A high total score indicates a high degree of catastrophizing pain.
Australian Pelvic Floor Questionnaire | Before and after eight weeks of vaginal surgery
  The Turkish version of the APFQ was shown to be valid and reliable. The scale assessing pelvic floor function has subheadings of bladder, bowel, prolapse, and sexual function. The total score ranges from 0-40. The high score indicates that severity of symptoms is high and poor sexual function.
Female Sexual Function Index | Before and after eight weeks of vaginal surgery
  FSFI was developed to assess sexual function in women. It was shown to be reliable and valid in Turkish with 19 questions. There are six sub-dimensions of sexual function: desire, arousal, lubrication, orgasm, satisfaction, and pain. Each item is scored on a 0-5 scale. An increase in the total score indicates an improvement in sexual function; an increase in the score in the pain parameter indicates a decrease in pain sensation. The scale score ranges from 2-36. The cut-off value is 26.5 to define sexual dysfunction.
Visual Analog Scale | Before and first day after surgery
  Post-operative pain intensity during urination and defecation will be assessed with a 0-10 cm VAS before discharge. Duration of pain and factors that increased and decreased pain will recorded. The duration of first micturition, defecation, and first passing gas in the postoperative period will recorded.

REFERENCES:
- [Result] Sariibrahim Astepe B, Koleli I. Translation, cultural adaptation, and validation of Australian pelvic floor questionnaire in a Turkish population. Eur J Obstet Gynecol Reprod Biol. 2019 Mar;234:71-74. doi: 10.1016/j.ejogrb.2019.01.004. Epub 2019 Jan 14. PMID 30665079
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] https://doi.org/10.1080/24750573.2017.1322672
- [Result] Horn-Hofmann C, Scheel J, Dimova V, Parthum A, Carbon R, Griessinger N, Sittl R, Lautenbacher S. Prediction of persistent post-operative pain: Pain-specific psychological variables compared with acute post-operative pain and general psychological variables. Eur J Pain. 2018 Jan;22(1):191-202. doi: 10.1002/ejp.1115. Epub 2017 Sep 20. PMID 28940665
- [Result] Lautenbacher S, Huber C, Kunz M, Parthum A, Weber PG, Griessinger N, Sittl R. Hypervigilance as predictor of postoperative acute pain: its predictive potency compared with experimental pain sensitivity, cortisol reactivity, and affective state. Clin J Pain. 2009 Feb;25(2):92-100. doi: 10.1097/AJP.0b013e3181850dce. PMID 19333152
- [Result] Ghezzi F, Uccella S, Cromi A, Siesto G, Serati M, Bogani G, Bolis P. Postoperative pain after laparoscopic and vaginal hysterectomy for benign gynecologic disease: a randomized trial. Am J Obstet Gynecol. 2010 Aug;203(2):118.e1-8. doi: 10.1016/j.ajog.2010.04.026. Epub 2010 Jun 3. PMID 20522410
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30665079/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/10782451/